CLINICAL TRIAL: NCT04240717
Title: Shared Decision Making on Immunotherapy in Oncology - Prospective, Randomized, Controlled Trial
Brief Title: Shared Decision Making on Immunotherapy in Oncology
Acronym: PEF-Immun
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Collaborators: Innovationsfonds des Gemeinsamen Bundesausschusses, Germany (Unknown)
Responsible Party: Principal Investigator, Christiane Bieber, Prof. Dr. med., Heidelberg University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01VSF18047
Record Dates: First submitted 2019-12-23; First posted 2020-01-27 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Patient Decision Aid; Treatment As Usual
Keywords: Shared Decision Making; Patient Empowerment; Immunotherapy; Melanoma; Patient Decision Aid
MeSH Terms: conditions — Patient Participation; Melanoma | interventions — Decision Support Techniques

STUDY DESIGN:
Intervention Model Description: Participants are assigned to the interventional group (decision aid) or the control group (treatment-as-usual).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient Decision Aid (Experimental): Patients review an interactive, web-based Patient Decision Aid regarding their treatment options. Afterwards they receive medical consultation.
  Interventions: Behavioral: Patient Decision Aid
- Treatment As Usual (No Intervention): Patients receive medical consultation.

INTERVENTIONS:
Behavioral: Patient Decision Aid — The Patient Decision Aid is an interactive, web-based tool that provides information on advanced melanoma and its treatment options with a strong focus on immunotherapies (i.e. response to therapy, risk of side effects).
  Other Names: Decision Aid
  Arms: Patient Decision Aid

SUMMARY:
Patients with advanced melanoma are confronted with a serious treatment decision. The current guideline recommends considering the option of immunotherapy with checkpoint inhibitors. The substances approved for this purpose differ greatly in their efficacy and the risk for adverse events. Besides, in about half of the patients with advanced melanoma a BRAF V600 Mutation is found. In these patients, in addition to immunotherapy, treatment with BRAF/MEK inhibitors must be considered.

Research on shared decision making suggests that patients achieve greater satisfaction with the decision if they are actively being involved in the decision-making process. To enable them to do so, an interactive, web-based patient decision aid (PtDA) informing about the treatment options for advanced melanoma will be developed and evaluated in a bicentric, prospective randomized controlled clinical trial.

The use of PtDA is expected to lead to a higher level of information about the benefits and risks of the various treatment options (primary hypothesis).

DETAILED DESCRIPTION:
Immunotherapies are regarded as a new, promising treatment option for patients with advanced melanoma. However, immunotherapies can cause massive up to life-threatening side effects. The risks and benefits vary considerably between the possible therapy options. Besides, in about half of the patients with advanced melanoma a BRAF V600 Mutation is found. In these patients, in addition to immunotherapy, treatment with BRAF/MEK inhibitors must be considered. This treatment option usually produces a rapid response. In most cases, however, melanomas develop resistance after about 12 months.

Therefore, patients with advanced melanoma and their treating physicians are confronted with a very complex and preference-sensitive decision situation. Support in the form of a Patient Decision Aid (PtDA) can be helpful to support this complex decision-making process.

In the first project phase, an interactive web-based PtDA on treatment options for advanced melanomas will be developed. In the second phase of the project, the PtDA will be evaluated in a prospective randomized controlled clinical trial. Patients with a diagnosis of advanced melanoma will be recruited at the National Center for Tumor Diseases (NCT) Heidelberg and at the University Cancer Center (UCC) Dresden.

Patients of the intervention group will receive access to the interactive PtDA prior to a medical consultation. Patients of the control group will receive the medical consultation only (treatment-as-usual). Group differences between the intervention group and the control group are analysed at T1 (immediately after the medical consultation) and T2 (three months after the medical consultation). The following variables are measured: informedness of the decision (primary outcome), decision satisfaction, and involvement of the patients in the decision process.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of metastatic melanoma (C43), stage 3 and 4
* first-line therapy
* tumor or metastases are not resectable
* sufficient knowledge of the German language to use the PtDA
* informed written consent to participate in the study

Exclusion Criteria:

* limited legal capacity or impairments in this respect
* cognitive or physical impairments, which severely complicate the use of the Patient Decision Aid (e.g. impaired vision)
* severe psychiatric or mental illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2020-02-07 (Actual); Primary Completion 2022-06-24 (Actual); Study Completion 2022-10-08 (Actual)

PRIMARY OUTCOMES:
Knowledge about different treatment options | T1 = after intervention (PtDA/TAU); duration of assessment: 10 minutes
  Knowledge is assessed by a self-developed multiple choice test assessing knowledge about course, benefits, risks, and mechanisms of actions of different treatment options. Higher scores indicate higher knowledge about treatment options.

SECONDARY OUTCOMES:
Decision satisfaction | T1 = after intervention (PtDA/TAU); duration of assessment: 2 minutes
  Decision satisfaction is assessed by the Satisfaction with Decision Scale (SwD; min. value: 6, max. value: 30; higher scores indicate higher satisfaction with decision)
Decision satisfaction (follow-up) | T2 = approx. 3 months after intervention (PtDA/TAU), before and after being informed about potential tumor progress; duration of assessment: 2 minutes
  Decision satisfaction is assessed with the same scale used at T1 (see Outcome 2 for a detailed description)
Patient involvement in the decision making process | during medical consultation; duration of assessment: approx. 30 minutes
  Patient involvement in the decision making process is assessed by the Observer OPTION 5 (min. value: 0, max. value: 20, higher scores indicate higher patient involvement in the decision making process)
Choice of treatment option | T1 = after the intervention (PtDA/TAU); duration of assessment: 1 minute
  Choice of treatment option is assessed by a self-developed item
Quality of physician-patient interaction | T1 = after the intervention (PtDA/TAU); duration of assessment: 2 minutes
  Quality of physician-patient interaction is assessed by the Questionnaire on the Quality of Physician-Patient Interaction (QQPPI, min. value: 14, max. value: 70, higher values indicate higher quality of physician-patient interaction)
Knowledge about different treatment options (follow-up) | T2: approx. 3 months after intervention (PtDA/TAU), before being informed about potential tumor progress; duration of assessment: 10 minutes
  Knowledge is assessed with the same multiple choice test used at T1 (see Outcome 1 for a detailed description).

CONTACTS AND LOCATIONS:
Overall Officials: Christiane Bieber, Prof. Dr., Principal Investigator — Heidelberg University
Locations (2):
- Germany (2):
  - University Hospital Heidelberg, Heidelberg, Baden-Wurttemberg
  - Carl Gustav Carus University Hospital Dresden, Dresden, Saxony

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Larkin J, Chiarion-Sileni V, Gonzalez R, Grob JJ, Rutkowski P, Lao CD, Cowey CL, Schadendorf D, Wagstaff J, Dummer R, Ferrucci PF, Smylie M, Hogg D, Hill A, Marquez-Rodas I, Haanen J, Guidoboni M, Maio M, Schoffski P, Carlino MS, Lebbe C, McArthur G, Ascierto PA, Daniels GA, Long GV, Bastholt L, Rizzo JI, Balogh A, Moshyk A, Hodi FS, Wolchok JD. Five-Year Survival with Combined Nivolumab and Ipilimumab in Advanced Melanoma. N Engl J Med. 2019 Oct 17;381(16):1535-1546. doi: 10.1056/NEJMoa1910836. Epub 2019 Sep 28. PMID 31562797
- [Background] Stacey D, Legare F, Lewis K, Barry MJ, Bennett CL, Eden KB, Holmes-Rovner M, Llewellyn-Thomas H, Lyddiatt A, Thomson R, Trevena L. Decision aids for people facing health treatment or screening decisions. Cochrane Database Syst Rev. 2017 Apr 12;4(4):CD001431. doi: 10.1002/14651858.CD001431.pub5. PMID 28402085
- [Background] Volk RJ, Llewellyn-Thomas H, Stacey D, Elwyn G. Ten years of the International Patient Decision Aid Standards Collaboration: evolution of the core dimensions for assessing the quality of patient decision aids. BMC Med Inform Decis Mak. 2013;13 Suppl 2(Suppl 2):S1. doi: 10.1186/1472-6947-13-S2-S1. Epub 2013 Nov 29. PMID 24624947
- [Background] Schadendorf D, van Akkooi ACJ, Berking C, Griewank KG, Gutzmer R, Hauschild A, Stang A, Roesch A, Ugurel S. Melanoma. Lancet. 2018 Sep 15;392(10151):971-984. doi: 10.1016/S0140-6736(18)31559-9. PMID 30238891
- [Derived] Grabbe P, Gschwendtner KM, Maatouk I, Strobel SB, Salzmann M, Bossert J, Eich W, Wild B, Meier F, Hassel JC, Bieber C. Development and validation of a web-based patient decision aid for immunotherapy for patients with metastatic melanoma: study protocol for a multicenter randomized trial. Trials. 2021 Apr 20;22(1):294. doi: 10.1186/s13063-021-05234-4. PMID 33879219